CLINICAL TRIAL: NCT04613453
Title: Reducing Adolescent Suicide Risk: Safety, Efficacy, and Connectome Phenotypes of Intravenous Ketamine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early due to concerns from the NIH DSMB regarding the rate of recruitment and the resulting inability to accomplish the initially approved study aims
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Bloch, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000029003; 1R01MH125203-01 (NIH)
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Adolescent Suicide; Adolescent Depression
Keywords: Intravenous Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine Infusion (Experimental): Participants will receive four Ketamine infusions over two weeks, each 0.5mg/kg over 40 minutes.
  Interventions: Drug: Ketamine Infusion
- Midazolam Infusion (Active Comparator): Participants will receive four Midazolam infusions over two weeks, each 0.045mg/kg over 40 minutes.
  Interventions: Drug: Midazolam Infusion

INTERVENTIONS:
Drug: Ketamine Infusion — Participants will receive four Ketamine infusions over two weeks, each 0.5mg/kg over 40 minutes.
  Arms: Ketamine Infusion
Drug: Midazolam Infusion — Participants will receive four Midazolam infusions over two weeks, each 0.045mg/kg over 40 minutes.
  Arms: Midazolam Infusion

SUMMARY:
The purpose of this study is to determine if intravenous ketamine reduces suicidal thinking compared to an active placebo (midazolam) in adolescents who have treatment resistant depression and a recent history of a suicide event (defined as a suicide attempt, emergency room evaluation for suicidal thinking, or a transition to inpatient care for suicidality in the past 120 days).

The primary objective of this study is to determine whether ketamine reduces suicidal ideation (as measured via the C-SSRS, recent ideation scale) relative to an active control, midazolam, 48-hours after first administration in adolescents with TRD at high suicide risk.

DETAILED DESCRIPTION:
The main purpose of the study is to examine the safety, efficacy, response predictors, and post-treatment trajectory of adolescents with TRD and high suicide risk following a highly conservative repeat dosing ketamine infusion paradigm (four infusions of 0.5mg/kg each over two weeks) compared to an active control, midazolam. Those who are randomized to midazolam and remain ill have the option to cross-over to ketamine in the open phase. All participants will be followed closely for four months post-treatment and treated with standard of care depression treatment (medication management and cognitive behavioral therapy). Brain-based predictors of anti-suicidal responses will be assessed via connectome predictive modeling (CPM), examining functional brain circuits via fMRI before and after treatment.

Given the unregulated use of ketamine in the community at widely varying doses and frequencies, the safety data gathered from this highly conservative repeat dosing paradigm is critical to inform the field about potential risks. Efficacy data at rapid, short-term, and intermediate-term (4 month) timepoints will be critical to determining whether a larger study is warranted in this population. The assessment of brain-based predictors of response through the integration of functional neuroimaging adds an important measure of biological engagement that will inform subsequent studies and stands to contribute towards the goal of personalized medicine (i.e. determining not only if a treatment works, but in whom).

Aim 1: To evaluate the safety of treating adolescents with TRD at high suicide risk with a conservative repeat-dosing ketamine paradigm followed by standard of care treatment over 4 months. Hypothesis: We anticipate no untoward effects on medical outcomes (cardiovascular function and bladder health) or cognitive function (measured via Cogstate).

Aim 2: To evaluate the 48-hour impact of ketamine on suicidal ideation compared to midazolam, and to identify connectome phenotypes predictive of ideation post-treatment. Hypothesis: Ketamine will reduce suicidal thinking (Columbia Suicide Rating Scale, recent ideation subscale) compared to midazolam. CPM will identify networks predictive of ideation, validated via k-fold or leave-one-out cross-validation within the sample. The network measures obtained at this fixed ketamine dose will inform the design of larger clinical trials.

Aim 3 (exploratory): To describe the trajectory of suicidal thinking, depressive symptoms, and use of mental health resources in both ketamine responders and non-responders over 4 months.

In July of this year (2024), the NIMH DSMB determined that Study 2000029003 will not be able to enroll enough individuals to be sufficiently powered to test the efficacy of Ketamine in treating adolescents with Major Depressive Disorder (MDD) and suicidal ideation (the primary aim of the study). Subsequently, the study was closed to enrollment

ELIGIBILITY:
Inclusion Criteria:

1. Ages 13-17 years, inclusive
2. Meet DSM-5 criteria for Major Depressive Disorder by structured interview (MINI-KID+)
3. Children's Depression Rating Scale, Revised (CDRS-R) score ≥45 at screening
4. Continued clinically significant depressive symptoms despite an SRI trial (e.g. SSRI or SNRI) of adequate dose and duration, meaning at least 6 weeks at therapeutic dosing, including at least 4 weeks of stable dosing
5. Suicide event within the past 120 days (i.e. a suicide attempt (defined as an act of potentially self-injurious behavior with explicit or inferred intent to die) -OR- degree of suicidal ideation requiring an emergency evaluation or a transition to higher level of care (e.g. intensive outpatient program, partial hospital program, inpatient)
6. Columbia Suicide Severity Rating Scale ideation score of ≥ 1 at screening
7. Medically and neurologically healthy on the basis of physical examination, medical history, and the clinical judgement of the evaluating physician.
8. Parents able to provide written informed permission and adolescents must additionally provide assent.
9. Stated willingness to comply with all study procedures and availability for the duration of the study
10. Provision of signed and dated parental permission and adolescent assent form. If there are two parents or guardians, both must provide permission and each must sign a separate permission form.

Exclusion Criteria:

1. History of psychotic disorder, manic episode, or autism spectrum disorder diagnosed by MINI-KID
2. History of substance dependence diagnosis by MINI-KID (excluding tobacco) or positive urine toxicology
3. Intellectual disability (IQ<70) per medical history
4. Pregnancy (urine pregnancy tests on the day of infusions for menstruating girls) or lactation
5. Prior participation in a ketamine study, prior clinical psychiatric treatment with ketamine, or prior recreational use of ketamine
6. Pre-existing cardiovascular disease or untreated or unstable hypertension
7. Body weight greater than 80 kgs
8. Currently taking benzodiazepines or other medications that may cause respiratory depression, or lamotrigine, which is hypothesized to interfere with ketamine's mechanism of action
9. Inability to provide written informed consent according to the Yale Human Investigation Committee (HIC) guidelines in English.

   For participation in the fMRI scans only (participants with contraindications to fMRI may still participate in all other portions of the trial, providing they meet all other inclusion/exclusion criteria):
10. Any contraindication to MRI including severe claustrophobia, or metal in the body (including mental dental braces)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bloch, MD MS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Last enrolled patient skipped the blinded phase and received open-label Ketamine.
Period: Blinded Phase
Arm/Group | Ketamine Infusion | Midazolam Infusion
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Open Phase
Arm/Group | Ketamine Infusion | Midazolam Infusion
Started | 6 | 6
Completed | 6 | 2
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Population: One participant who was consented but not randomized at the time of study termination was offered unblinded ketamine and was included in the safety data for ketamine for the overall sample but not the efficacy analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Infusion | Midazolam Infusion | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 11
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1 | 1 | 2
  Female | 4 | 4 | 8
  Non-binary | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 6 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 5 | 8
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11
Age of depression onset [Median (Inter-Quartile Range); unit: years] | 13 [12 to 13] | 12 [11 to 15] | 12.5 [11 to 14]
Screening Children's Depression Rating Scale-Revised (CDRS-R) [Median (Inter-Quartile Range); unit: score on a scale] — CDRS-R is a 17-item scale examines depressive symptoms in children and adolescents using the combined report of the adolescent and the parent, synthesized by a clinician. This 17-item clinical scale creates scores that range from 17 to 113, with higher scores representing more intensive depressive symptoms
  score on a scale | 65.5 [65 to 68] | 75 [69 to 86] | 68.5 [65 to 78]
Screening Columbia-Suicide Severity Rating Scale (C-SSRS) [Median (Inter-Quartile Range); unit: score on a scale] — The C-SSRS is an assessment of suicidal ideation and behavior in clinical and research settings. The C-SSRS consists of 16 questions that ask about suicidal ideation and behaviors. This 5-item subscale ranges from a minimum of 0 (corresponding to no suicidal ideation) to a maximum of 5 (representing active suicidal ideation with plan and intent).
  score on a scale | 5 [4 to 5] | 5 [4 to 5] | 5 [4 to 5]
Number of previous antidepressant trials [Median (Inter-Quartile Range); unit: trials] | 3 [2 to 4] | 3.5 [2 to 4] | 3 [2 to 4]
Number of prior suicide attempts [Median (Inter-Quartile Range); unit: suicide attempts] | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 2.5]
Number of participants with Co-morbid anxiety disorder [Count of Participants; unit: Participants] | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is an assessment of suicidal ideation and behavior in clinical and research settings. The C-SSRS consists of 16 questions that ask about suicidal ideation and behaviors (the first 10 questions comprise the ideation subscale and the last 6 comprise the behavior subscale). Total score ranges for suicidal ideation from a minimum of 0 (corresponding to no suicidal ideation) to a maximum of 5 (representing active suicidal ideation with plan and intent). Total score ranges for suicidal behavior from a minimum of 0 (corresponding to no suicidal behavior) to a maximum of 5 (representing active suicidal behavior).
Time Frame: Baseline and Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Infusion | Midazolam Infusion
Number analyzed (Participants) | 5 | 6
score on a scale
  Baseline Suicidal Ideation | 2.60 (1.34) | 2.67 (1.37)
  Day 3 Suicidal Ideation | 1.20 (1.10) | 1.17 (1.60)
  Baseline Suicidal Behavior | 0.20 (0.45) | 0.41 (0.45)
  Day 3 Suicidal Behavior | 0 (0) | 0 (0)

2. Secondary Outcome: Montgomery Asberg Depression Rating Scale
Description: Montgomery Asberg Depression Rating Scale is an 10-item scale examines depressive symptoms and will be assessed at baseline (prior to any experimental treatment), prior to each experimental treatment, and weekly during the open phase of the trial. This 10-item scale ranges from 0 to 60, with higher values representing more intensive depressive symptoms.
Time Frame: Baseline and Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Infusion | Midazolam Infusion
Number analyzed (Participants) | 5 | 6
score on a scale
  Baseline | 30.4 (2.07) | 33 (11.93)
  Day 3 | 27.2 (4.44) | 24.17 (17.57)

3. Secondary Outcome: Change in Children's Depression Rating Scale
Description: Children's Depression Rating Scale-Revised is a 17-item scale examines depressive symptoms in children and adolescents using the combined report of the adolescent and the parent, synthesized by a clinician. It will be administered at baseline (prior to any experimental treatment), at the end of the blinded phase of the trial (Day 11), and monthly during the open phase of the trial. This 17-item clinical scale creates scores that range from 17 to 113, with higher scores representing more intensive depressive symptoms
Time Frame: Baseline to Day 11
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ketamine Infusion | Midazolam Infusion
Number analyzed (Participants) | 5 | 6
score on a scale
  Baseline | 69.5 [61 to 75] | 68 [59 to 84]
  Day 11 | 54.5 [42 to 71] | 66 [58 to 73]

ADVERSE EVENTS:
Time Frame: 4 months
Groups:
- Ketamine Infusion-Blinded: Participants will receive four Ketamine infusions over two weeks, each 0.5mg/kg over 40 minutes.
- Midazolam Infusion-Blinded: Participants will receive four Midazolam infusions over two weeks, each 0.045mg/kg over 40 minutes.
- Ketamine Infusion-Unblinded: 5 of 6 participants did not respond to Midazolam and received Ketamine infusions over two weeks, each 0.5mg/kg over 40 minutes as per protocol.
Arm/Group | Ketamine Infusion-Blinded | Midazolam Infusion-Blinded | Ketamine Infusion-Unblinded
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/5 | 3/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/5 | 5/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine Infusion-Blinded (N=5) | Midazolam Infusion-Blinded (N=6) | Ketamine Infusion-Unblinded (N=6)
Emergency Department Visit (General disorders) | 1 | 0 | 0
Self harm (Psychiatric disorders) | 2 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine Infusion-Blinded (N=5) | Midazolam Infusion-Blinded (N=6) | Ketamine Infusion-Unblinded (N=6)
Vision blurred (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Fatigue (General disorders) | 1 | 3 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 4
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Sedation (Nervous system disorders) | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 4 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 2
Asthenia (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Illusion (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Self-destructive behaviour (Psychiatric disorders) | 0 | 3 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Menstrual discomfort (Reproductive system and breast disorders) | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0
Atypical Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Skin hemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT04613453/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT04613453/ICF_001.pdf